CLINICAL TRIAL: NCT03550547
Title: Evaluation of the Added Value of an Educational Program Associated With a Conventional Spa Therapy of Knee Osteoarthritis Patients
Brief Title: Educational Program Associated With a Conventional Spa Therapy of Knee Osteoarthritis Patients
Acronym: GETT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A03323-50
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Knee Osteoarthritis
Keywords: Physical Activity; Education; Dietary; Self-management
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7 educational workshops (Experimental): Intervention: 7 educational workshops in addition to spa therapy :
  Knowledge of the pathology ; Educational physical activity ( 2 workshops); Dietary; Management of pain, fatigue and the medical treatments; Articular hygiene and ergonomics; Technical assistance, an adaptation of the living condition
  Interventions: Other: Educational workshops; Other: Spa Therapy
- spa therapy (Active Comparator): Approved Spa therapy
  Interventions: Other: Spa Therapy

INTERVENTIONS:
Other: Educational workshops — 1 workshop : Knowledge of the pathology ; 2a workshop: Educational physical activity; 2b workshop : Educational physical activity; 4 workshop : Dietary; 5 workshop : Management of pain, fatigue and the medical treatments; 6 workshop : Articular hygiene and ergonomics; 7 workshop : Technical assistance, an adaptation of the living condition
  Other Names: Non pharmacological intervention
  Arms: 7 educational workshops
Other: Spa Therapy — Approved Spa therapy of knee osteoarthritis patients
  Other Names: Non pharmacological intervention

SUMMARY:
The main objective of this work is to measure the efficiency of 18 days SPA Therapy in orientation rheumatology associated with an educational intervention in patients with knee osteoarthritis on a priority objective, personalized and determined by the patient, chosen in the list of 5 objectives determined during the educational assessment.

DETAILED DESCRIPTION:
This program begin with a shared educational balance assessment allowing to set up the individual program adapted to the objectives personalized by the patients. The objectives to achieve are to allow the patients to acquire knowledge and skills (attitudes, behavior) concerning their pathology and the existing treatment. A multidisciplinary team trained in the therapeutic education of the patient assure the educational interventions. The proposed educational activities (7 educational workshops) concern major axes of the care of the knee osteoarthritis: knowledge of the pathology, the adapted physical exercise, the dietetics, the management of the pain, the articular hygiene and the technical helps.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, aged 50 to 75 years
* Patients with knee osteoarthritis clinical criteria of the American College of Rheumatology (ACR)
* Patient affiliated to a social security scheme (beneficiary entitled)
* Patient registered spa
* Pain intensity equal or more than "3" at the Visual Analogical Scale
* Patient has given its consent in writing to

Exclusion Criteria:

* Contraindication to the spa therapy
* Trouble behavior or understanding making it impossible to assess

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-11-28 (Estimated); Study Completion 2022-05-28 (Estimated)

PRIMARY OUTCOMES:
Measuring effectiveness of the educational workshops, personalized and determined for every patient. | Month 06
  Average change from effectiveness of the educational workshops, personalized and determined for every patient, measured by a GAS GAS (Goal Attainment Scaling in Rehabilitation) is a method of scoring the extent to which patient's individual goals are achieved in the course of intervention. In effect, each patient has their own outcome measure but this is scored in a standardized way as to allow statistical analysis.
  Each goal is rated on a 5-point scale, with the degree of attainment captured for each goal area:
  * If the patient achieves the expected level, this is scored at 0.
  * If they achieve a better than expected outcome this is scored at: +1 (more than expected), +2 (much more than expected)
  * If they achieve a worse than expected outcome this is scored at: -1 (less than expected) or -2 (much less than expected) GAS depends on two things - the patient's ability to achieve their goals and the clinician's ability to predict outcome, which requires knowledge and experience.

SECONDARY OUTCOMES:
Functional status | Day 01, Day 18, Month 03, Month 06, Month 09, Month 12.
  Score on WOMAC
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items), stiffness (2 items), physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Pain intensity | Day 01, Day 18, Month 03, Month 06, Month 09, Month 12.
  Average change from baseline in the pain intensity measured on a Visual Analogical Scale (VAS) Visual analog scale (VAS) and its corresponding visual analog pain scale, is a psychometric scale that is generally used to conduct pain scale surveys to understand varying degrees of pain or discomfort experienced by a patient. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
Life quality | Day 01, Day 18, Month 03, Month 06, Month 09, Month 12.
  Average change from baseline of the Life quality, measured by a SF36. It is one of the most widely used generic measures of health-related quality of life and has been shown to discriminate between subjects with different chronic conditions and between subjects with different severity levels of the same disease. The SF-36 has also demonstrated sensitivity to significant treatment effects in a variety of patient populations. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Comprehensive evaluation of patient education programs | Day 18, Month 03, Month 06, Month 09, Month 12
  Average change from baseline of the comprehensive evaluation of patient education programs , measured by a HEIQ.
  The Health Education Impact Questionnaire (heiQ): an outcomes and evaluation measure for patient education and self-management interventions for people with chronic conditions.
  There are 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section, i.e. if one question is scored 1 and another 2, then the score for the section is 2.
Measuring effectiveness of the educational workshops, personalized and determined for every patient. | Day 01, Day 18, Month 03, Month 09, Month 12.
  Average change from effectiveness of the educational workshops, personalized and determined for every patient, measured by a GAS
  GAS (Goal Attainment Scaling in Rehabilitation) is a method of scoring the extent to which patient's individual goals are achieved in the course of intervention. In effect, each patient has their own outcome measure but this is scored in a standardized way as to allow statistical analysis.
  Each goal is rated on a 5-point scale, with the degree of attainment captured for each goal area:
  * If the patient achieves the expected level, this is scored at 0.
  * If they achieve a better than expected outcome this is scored at: +1 (more than expected), +2 (much more than expected)
  * If they achieve a worse than expected outcome this is scored at: -1 (less than expected) or -2 (much less than expected) GAS depends on two things - the patient's ability to achieve their goals and the clinician's ability to predict outcome, which requires knowledge and experience.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, MD-PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Etablissement thermal, Dax, Aquitaine, France

REFERENCES:
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131
- [Background] Mendelson AD, McCullough C, Chan A. Integrating self-management and exercise for people living with arthritis. Health Educ Res. 2011 Feb;26(1):167-77. doi: 10.1093/her/cyq077. Epub 2010 Dec 1. PMID 21123844
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Krasny-Pacini A, Evans J, Sohlberg MM, Chevignard M. Proposed Criteria for Appraising Goal Attainment Scales Used as Outcome Measures in Rehabilitation Research. Arch Phys Med Rehabil. 2016 Jan;97(1):157-70. doi: 10.1016/j.apmr.2015.08.424. Epub 2015 Sep 4. PMID 26343173
- [Background] Rockwood K, Joyce B, Stolee P. Use of goal attainment scaling in measuring clinically important change in cognitive rehabilitation patients. J Clin Epidemiol. 1997 May;50(5):581-8. doi: 10.1016/s0895-4356(97)00014-0. PMID 9180650
- [Derived] Goldstein A, Lanhers C, Gay C, Dubourg K, Grange L, Roques CF, Pereira B, Coudeyre E. Efficacy of self-management program associated with a spa therapy for knee osteoarthritis patients (GETT 2): a research protocol for a randomized trial. Trials. 2023 Jan 19;24(1):45. doi: 10.1186/s13063-022-06879-5. PMID 36658607